CLINICAL TRIAL: NCT05929469
Title: PATH to Health: An Exploration of Digital Behavioral Weight Loss Approaches
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Academy of Nutrition and Dietetics (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 23-0396
Record Dates: First submitted 2023-06-13; First posted 2023-07-03 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2023-10

CONDITIONS: Overweight; Obesity; Overweight and Obesity
Keywords: Behavioral intervention; SMART (sequential multiple assignment randomized trial)
MeSH Terms: conditions — Overweight; Obesity | interventions — Amyloid; Counseling

STUDY DESIGN:
Intervention Model Description: This initial pilot and feasibility study uses a sequential, multiple assignment, randomized trial (SMART) design to test digital, behavioral weight loss approaches, with or without human support. Sequential randomization will occur at baseline and at the end of 4 weeks. At baseline, participants will be randomized to receive a standard mHealth program and either a a) Fully Automated Kick-Off session, or b) Human-Enhanced Kick-Off session. Using an a priori decision rule after 4 weeks, those for whom the intervention is not effective will be re-randomized and receive one of two doses of human support. The final assessment will be at 3 months.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Fully Automated Kick-Off + App (Experimental): This arm includes participants who respond to the Fully Automated Kick-Off + App in stage 1.
  In stage 1, participants will receive a Fully Automated Kick-Off and an mHealth program.
  In stage 2, responders to the Fully Automated Kick-Off + App will continue with the mHealth program, alone, for the remainder of the study.
  Interventions: Behavioral: App; Behavioral: Fully Automated Kick-Off
- Human-Enhanced Kick-Off + App (Experimental): This arm includes participants who respond to the Human-Enhanced Kick-Off + App in stage 1.
  In stage 1, the participant's kick-off will include a session with a study interventionist. They will also receive an mHealth program.
  In stage 2, responders to the Human-Enhanced Kick-Off + App will continue with the mHealth program, alone, for the remainder of the study.
  Interventions: Behavioral: App; Behavioral: Human-Enhanced Kick-Off
- Fully Automated Kick-Off + App + Check-In (Experimental): This arm includes participants who do not respond to the Fully Automated Kick-Off + App in stage 1.
  In stage 1, participants will receive a Fully Automated Kick-Off and an mHealth program.
  In stage 2, they will continue with the mHealth program, but will also receive a check-in with a study interventionist.
  Interventions: Behavioral: App; Behavioral: Fully Automated Kick-Off; Behavioral: Check-In
- Fully Automated Kick-Off + App + Counseling (Experimental): This arm includes participants who do not respond to the Fully Automated Kick-Off + App in stage 1.
  In stage 1, participants will receive a Fully Automated Kick-Off and an mHealth program.
  In stage 2, they will continue with the standard mHealth program, but will also receive counseling from a study interventionist.
  Interventions: Behavioral: App; Behavioral: Fully Automated Kick-Off; Behavioral: Counseling
- Human-Enhanced Kick-Off + App + Check-In (Experimental): This arm includes participants who do not respond to the Human-Enhanced Kick-Off + App in stage 1.
  In stage 1, the participant's kick-off will include a session with a study interventionist. They will also receive an mHealth program.
  In stage 2, they will continue with the mHealth program, but will also receive a check-in with a study interventionist.
  Interventions: Behavioral: App; Behavioral: Human-Enhanced Kick-Off; Behavioral: Check-In
- Human-Enhanced Kick-Off + App + Counseling (Experimental): This arm includes participants who do not respond to the Human-Enhanced Kick-Off + App in stage 1.
  In stage 1, the participant's kick-off will include a session with a study interventionist. They will also receive an mHealth program.
  In stage 2, they will continue with the standard mHealth program, but will also receive counseling from a study interventionist.
  Interventions: Behavioral: App; Behavioral: Human-Enhanced Kick-Off; Behavioral: Counseling

INTERVENTIONS:
Behavioral: App — Participants will receive an mHealth program.
Behavioral: Fully Automated Kick-Off — As an orientation to the study, participants will receive a fully automated kick-off session.
  Arms: Fully Automated Kick-Off + App; Fully Automated Kick-Off + App + Check-In; Fully Automated Kick-Off + App + Counseling
Behavioral: Human-Enhanced Kick-Off — As an orientation to the study, participants will receive a kick-off session that includes time with a study interventionist.
  Arms: Human-Enhanced Kick-Off + App; Human-Enhanced Kick-Off + App + Check-In; Human-Enhanced Kick-Off + App + Counseling
Behavioral: Check-In — Participants will receive a check-in with a study interventionist.
  Arms: Fully Automated Kick-Off + App + Check-In; Human-Enhanced Kick-Off + App + Check-In
Behavioral: Counseling — Participants will receive counseling from a study interventionist.
  Arms: Fully Automated Kick-Off + App + Counseling; Human-Enhanced Kick-Off + App + Counseling

SUMMARY:
The purpose of this initial pilot and feasibility study is to test different digital, behavioral weight loss approaches, with or without human support, using a sequential, multiple assignment, randomized trial (SMART) design. All participants in this pilot trial will receive a 3-month mobile health (mHealth) program. The dose of human support will vary by first- and second-line randomizations. The feasibility, acceptability, and preliminary outcomes for each of the treatment sequences will be assessed.

DETAILED DESCRIPTION:
Ninety-nine adults, ages 18-65, with overweight or obesity, will be randomized in total. All participants will receive an mHealth program (App) for program duration that includes activity tracking with a Fitbit, weight tracking with a smart scale, and an app for diet tracking. At baseline, participants will be randomized to either a a) Fully Automated Kick-Off, or b) Human-Enhanced Kick-Off. "Early responders" will continue with to use App, alone. After 4 weeks, "early non-responders" in both arms will be re-randomized once to one of two augmented interventions with human support: Counseling or Check-In. Assessments will occur at baseline, 1 week, 4 weeks, and 3 months to explore feasibility, acceptability, and preliminary outcomes (weight, self-monitoring adherence, behavioral goal adherence).

ELIGIBILITY:
Inclusion Criteria:

* Current age: 18-65 years
* Lives in North Carolina
* Body mass index (BMI) of 27.5-45 kg/m^2
* Ability to read, write, and speak English
* Ownership of iPhone with a data and texting plan
* Ability to commit to the required counseling sessions (0-5 sessions, based on randomization)
* Is not living a participant or staff member on this trial
* Willingness to be randomized to any of the treatment sequences

Exclusion Criteria:

* Weight loss of more than 10 pounds in the last 6 months that was maintained
* A history of weight loss surgery
* Pre-existing medical condition(s) that prevent them from adhering to a supervised exercise routine
* Have Type 1 Diabetes or are currently taking medicine for Type 2 Diabetes
* Have recently been diagnosed or treated for cancer
* Currently pregnant, pregnant within the past 6 months, or plan to become pregnant in the next 6 months
* Report taking prescription or over the counter medication with a known impact on metabolism or weight
* Report a history of an eating disorder
* History of psychotic disorder or bipolar disorder, or have been hospitalized for depression or other psychiatric disorder within the past 12 months
* History of alcohol or substance abuse
* Current participation in another weight loss program that may interfere with participation in this study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2023-10-02 (Actual); Primary Completion 2024-04-25 (Actual); Study Completion 2024-04-25 (Actual)

PRIMARY OUTCOMES:
Feasibility- Rate of early nonresponse | 4 weeks
  The rate of early response will be calculated as the number of individuals deemed "early responders" divided by the total number of participants randomized.
Feasibility- Percentage of participants with missing data at 4 weeks | 4 weeks
  The percentage of participants with missing data at 4 weeks will be calculated as the number of participants who do not complete the 4-week weight assessment divided by the total number of participants randomized.

SECONDARY OUTCOMES:
Weight Change- Percent weight change from baseline to 3 months | Baseline, 3 months
  Percent weight change from baseline to 3 months will be calculated ((3 month weight - baseline weight)/100). Weight will be objectively measured on a scale in the participant's home.
Weight Change- Percent weight change from baseline to 4 weeks | Baseline, 4 weeks
  Percent weight change from baseline to 4 weeks will be calculated ((4 week weight - baseline weight)/100). Weight will be objectively measured on a scale in the participant's home
Weight Change- Percent weight change from 4 weeks to 3 months | 4 weeks, 3 months
  Percent weight change from 4 weeks to 3 months will be calculated ((3 month weight - 4 week weight)/100). Weight will be objectively measured on a scale in the participant's home
Acceptability- Rate of attendance at human support sessions | Up to 3 months
  The rate of attendance at human support sessions will be calculated as the number of human sessions completed divided by the number of human sessions assigned.
Acceptability- Attrition | Up to 3 months
  Attrition will be calculated as the number of intervention participants who did not complete 3-month weight measures divided by the number randomized to treatment.
Acceptability- Overall program satisfaction rating | 3 months
  Overall program satisfaction will be assessed using a single item, which asks participants to rate their overall satisfaction with the program on a 4-point Likert scale that ranges from "very dissatisfied" to "very satisfied," in which higher scores indicate greater levels of satisfaction.
Weighing Self-Monitoring Adherence | Baseline to 3 months (daily)
  Number of days of self-weighing over the 3 month period, measured by use of the scale in the participant's home.
Dietary Self-Monitoring Adherence | Baseline to 3 months (daily)
  Number of days of complete dietary tracking summed over the 3-month study period, as measured by app use data.
Physical Activity Self-Monitoring Adherence | Baseline to 3 months (daily)
  Number of days of physical activity tracking over the 3 month period, as measured by Fitbit tracker wear.
Dietary Goal Adherence | Baseline to 3 months (daily)
  Number of days the participant met their daily calorie goal over the 3 month period, as measured by app data.
Activity Goal Adherence | Baseline to 3 months (daily)
  Number of days the participant met their active minutes goal over the 3 month period, as measured by app data.
Change in Diet | Baseline, 3 months
  Change in daily caloric intake from baseline to 3 months, as measured using the self- administered National Cancer Institute's Automated Self- Administered 24-hour Recall (ASA-24), a 24-hour recall that is self-administered on one day at each timepoint.
Change in Physical Activity | Baseline, 3 months
  Change in physical activity from baseline to 3 months, as measured using the Paffenbarger Physical Activity Questionnaire (PPAQ). The PPAQ assesses amount of planned and lifestyle associated physical activity performed during a typical week. The PPAQ consists of three components: (1) stair climbing, (2) walking, and (3) sports and recreation. Participants report the frequency and duration of physical activity in the past week. Scoring yields energy expenditure from physical activity per week (kcal/kg/week). Higher scores translate into greater energy expenditure per week (i.e.,better outcome). Range is 0 - no theoretical maximum.
Change in Motivation | Baseline, 1 week, 4 weeks, 3 months
  Change in motivation from baseline to 4 weeks and 3 months, as measured using the Treatment Self-Regulation Questionnaire (TSRQ). The TSRQ assesses autonomous and controlled motivation for weight management. Six items assess autonomous motivation and six assess controlled motivation using a 7 point Likert scale, in which 1 corresponds to "not at all true" and 7 corresponds to "very true." Items will be averaged to produce scores for autonomous motivation and controlled motivation ranging from 1-7. Higher values on each sub-scale indicate greater levels of that type of motivation. A Relative Autonomous Index (RAI) score will be separately calculated by subtracting the controlled motivation score from the autonomous motivation score. The range of possible RAI scores is -6 to 6.

CONTACTS AND LOCATIONS:
Overall Officials: Caitlin Martinez, MS, RD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Martinez CE, Nezami BT, Mayer-Davis E, Willis EA, Gorin AA, Tate DF. Results of a pilot sequential multiple assignment randomized trial using counseling to augment a digital weight loss program. Obes Sci Pract. 2024 Nov 7;10(6):e70018. doi: 10.1002/osp4.70018. eCollection 2024 Dec. PMID 39512729